CLINICAL TRIAL: NCT00657046
Title: A Phase II, Multi-center, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Assess the Clinical Benefit and Safety of Droxidopa in Patients With Intradialytic Hypotension
Brief Title: Safety and Benefit Study of Droxidopa to Treat Patients With Intradialytic Hypotension
Acronym: IDH201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Droxidopa IDH201
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Intradialytic Hypotension
MeSH Terms: interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Droxidopa at 400 mg (2 capsules each containing 200 mg droxidopa plus one capsule with Placebo)
  Interventions: Drug: Droxidopa; Drug: Placebo
- 2 (Active Comparator): Droxidopa at 600 mg (3 capsules each containing 200 mg droxidopa)
  Interventions: Drug: Droxidopa
- 3 (Placebo Comparator): Placebo (3 capsules with mannitol substituted for droxidopa)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Droxidopa — Capsules containing 200 mg droxidopa
  Arms: 1; 2
Drug: Placebo — Capsules with mannitol substituted for droxidopa
  Arms: 1; 3

SUMMARY:
In clinical trials in Japan, droxidopa has been shown to be effective in affecting blood pressure changes upon orthostatic challenge in patients with autonomic dysfunction, as well as reducing the severity and frequency of symptoms of orthostatic hypotension in these patients. The efficacy of droxidopa in ameliorating symptoms in patients undergoing dialysis has also been demonstrated in the literature and clinical trials conducted in Japan. The current study will investigate the clinical efficacy of two different doses of droxidopa in patients with intradialytic hypotension over a 4 week treatment period with a placebo control. The clinical efficacy will be evaluated by changes in hypotension- related symptoms, as well as changes in blood pressure prior to, during and following, HD sessions as compared to their pre-treatment baseline values.

DETAILED DESCRIPTION:
This is a phase II, multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of droxidopa in HD patients with intradialytic hypotension. The study will be conducted in up to 15 centers, with a sufficient number of patients enrolled to allow 75 patients to be randomized into 3 study groups (25 randomized to placebo, 25 randomized to 400 mg droxidopa, and 25 randomized to 600 mg droxidopa).

The study will consist of an initial screening period (up to 7 days) to confirm eligibility followed by a 2 week baseline, and a 4 week treatment period. During baseline and treatment visits SBP and DBP measurements will be collected using a consistent method immediately pre-, during and immediately post-dialysis. SBP, DBP and heart rate measurements will be taken every 20 minutes during HD sessions.

There will be 19 scheduled visits, not including the post-treatment follow-up visit, during this trial; Visit 1 (Screening), Visits 2 through 7 (baseline and randomization), Visits 8 through 19 (tri-weekly treatment visits). Each visit will coincide with the patient's normal dialysis treatments.

All patients will be followed for 30 days following the completion of the active treatment period (or premature withdrawal) to check for the occurrence of adverse events (AEs).

Patients will attend the study center as out-patients.

Eligible patients will be assigned a unique identification number at screening, and prior to the first treatment visit will be randomized to one of the following treatment groups:

Group A: Droxidopa at 400 mg (2 capsules each containing 200 mg droxidopa plus one capsule with mannitol substituted for droxidopa) Group B: Droxidopa at 600 mg (3 capsules each containing 200 mg droxidopa) Group C: Placebo (3 capsules with mannitol substituted for droxidopa) Each patient will take 3 capsules 1 hour prior to each dialysis procedure with approximately 100 mL (typically half a glass) of water.

The primary measure of efficacy will be the change from baseline (visits 2-7) in average mean arterial blood pressure compared to that during treatment (visit 14-19).

The secondary measures of efficacy will be:

* Change between baseline (visits 2-7) and treatment (visits 14-19) in average mean nadir systolic and diastolic blood pressures during hemodialysis;
* Change in the number of hypotension-induced interventions during hemodialysis (HD) sessions;
* Change in hypotension-induced symptoms measured during hemodialysis;
* Change in daily symptoms associated with hemodialysis;
* Change in fatigue using the Multidimensional Fatigue Inventory (MFI-20). The safety of droxidopa will be evaluated based on the occurrence of treatment-emergent adverse events (AE) and specific evaluation of blood pressure, heart rate (HR), ECG, and laboratory findings across the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and aged 18 years or over;
2. Clinical diagnosis of ESRD;
3. Demonstrated requirement to undergo maintenance HD 3 times per week for sessions at least 3 hours in duration;
4. Medical history consistent with IDH existing for at least 1 month;
5. Observed symptomatic intradialytic hypotension in 3 of 6 HD sessions during screening, as defined by as a decrease in systolic blood pressure by ≥20 mm Hg or a decrease in MAP by 10 mm Hg associated with symptoms that include: abdominal discomfort; yawning; sighing; nausea; vomiting; muscle cramps; restlessness; dizziness or fainting; and anxiety (definition according to: National Kidney Foundation 2007) ;
6. Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care.

Exclusion Criteria:

1. Currently taking ephedrine or midodrine;

   * Patients taking ephedrine or midodrine may enroll after a minimum 7 day washout period
2. Taking anti-hypertensive medication on the day of dialysis;
3. Currently taking selective norepinephrine re-uptake inhibitors;
4. Current known or suspected drug or substance abuse;
5. Women of childbearing potential who are not using a medically accepted contraception;

   Subject Restrictions:
   * Reproductive potential: Female subjects should be either post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile, or women of child-bearing potential (WOCP) who are using or agree to use acceptable methods of contraception. Acceptable contraceptives include intrauterine devices (IUDs), hormonal contraceptives (oral, depot, patch or injectable) and double barrier methods such as condoms or diaphragms with spermicidal gel or foam.
   * For WOCP a urine/serum beta HCG pregnancy test must be conducted at screening and study termination, and a urine/serum pregnancy test must be conducted at baseline; the results must be negative at screening and at baseline. WOCP must be advised to use acceptable contraceptives throughout the study period and for 30 days after the last dose of investigational product. If hormonal contraceptives are used they should be taken according to the package insert. WOCP who are not currently sexually active must agree to use acceptable contraception, as defined above, if they decide to become sexually active during the period of the study and for 30 days after the last dose of investigational product.
6. Sexually active males whose partner is a WOCP must agree to use condoms for the duration of the study and for 30 days after the last dose;
7. Women who are pregnant or breast feeding;
8. Known or suspected hypersensitivity to the study medication or any of its ingredients;
9. Have active atrial fibrillation (within the last 6 months) or, in the investigator's opinion, have any other significant cardiac arrhythmia;
10. Any other significant systemic, hepatic or cardiac illness;
11. Have a history of closed angle glaucoma;
12. Have a known or suspected malignancy (other than basal cell carcinoma);
13. Patients with known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug;
14. In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing;
15. In the investigator's opinion, are unable to adequately cooperate because of individual or family situation;
16. In the investigator's opinion, are suffering from a mental disorder that interferes with the diagnosis and/or with the conduct of the study, e.g. schizophrenia, major depression, dementia;
17. Are not able or willing to comply with the study requirements for the duration of the study;
18. Have participated in another clinical trial with an investigational agent (including named patient or compassionate use protocol) within 30 days before the start of the study;
19. Previous enrollment in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Halligan, MD, Principal Investigator — Bayview Nephrology
Locations (1):
- Rogue Valley Dialysis, Medford, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Droxidopa 400mg: Droxidopa at 400 mg (2 capsules each containing 200 mg droxidopa plus one capsule with mannitol substituted for droxidopa) taken 1 hour (+/-15 minutes) prior to each hemodialysis session. Study treatments were administered over 4 weeks.
- Droxidopa 600mg: Droxidopa at 600 mg (3 capsules each containing 200 mg droxidopa) taken 1 hour (+/-15 minutes) prior to each hemodialysis session. Study treatments were administered over 4 weeks.
- Placebo: Placebo (3 capsules with mannitol substituted for droxidopa) taken 1 hour (+/-15 minutes) prior to each hemodialysis session. Study treatments were administered over 4 weeks.
Period: Overall Study
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Started | 30 | 32 | 23
Had at Least 1 Post Baseline Visit | 30 | 31 | 23
Had Visits up to Visit 18 | 28 | 30 | 23
Completed | 26 | 29 | 21
Not Completed | 4 | 3 | 2
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Surgery | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 23 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (12.71) | 59.7 (14.98) | 60.2 (16.00) | 60.0 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 14 | 47
  Male | 14 | 15 | 9 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 15 | 12 | 46
  White | 11 | 17 | 11 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 32 | 23 | 85

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Mean Arterial Blood Pressure During Hemodialysis
Description: Change between average baseline (visits 2-7) mean arterial blood pressure during hemodialysis and average treatment (visits 14-19) mean arterial blood pressure during hemodialysis.
  The calculation of MAP was based on the systolic (SBP) and diastolic (DBP) blood pressure measurements taken during each valid HD session, using the traditional formula:
  MAP = (SBP+2*DBP)/3 for each time-point. The mean of the intradialytic measurements was calculated for each valid HD session, and these daily mean values were averaged across the visits within each period.
Time Frame: 6 weeks
Population: Patients must have blood pressure data from baseline and from visits 14-19. One droxidopa 400mg patient did not have blood pressure data for visit 14-19 and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 27 | 30 | 23
mmHg | -0.12 (10.017) | 1.95 (6.637) | 1.60 (9.843)
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.693, ANCOVA; GLM model with baseline as a covariate
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.807, ANCOVA; GLM model with baseline as a covariate

2. Secondary Outcome: Change in Average Mean Nadir Systolic Blood Pressures During Hemodialysis;
Description: Change between baseline (visits 2-7) and treatment (visits 14-19) in average mean nadir systolic blood pressures during hemodialysis. The baseline value will be the arithmetic average of the values collected at each of the six baseline visits (visits 2-7). The on treatment value will be defined as the average of the values collected at each of the last six treatment visits (visits 14-19).
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 27 | 30 | 23
mmHg | 3.09 (16.065) | 2.60 (9.988) | -0.35 (14.695)
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.212, ANCOVA; GLM model with baseline as a covariate
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.230, ANCOVA; GLM model with baseline as a covariate

3. Secondary Outcome: Change in the Number of Hypotension-induced Interventions During Hemodialysis (HD) Sessions;
Description: Evaluate the efficacy of droxidopa as measured by change in the number of hypotension-induced interventions during hemodialysis (HD) sessions between baseline (visits 2-7) and treatment (visits 14-19). The baseline value will be the arithmetic average of the values collected at each of the six baseline visits (visits 2-7). The on treatment value will be defined as the average of the values collected at each of the last six treatment visits (visits 14-19).
Time Frame: 6 weeks
Population: Patients must have completed visits in the visit 14-19 timeframe.
Measure: Mean (Standard Deviation); unit: average interventions per session
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 28 | 30 | 23
average interventions per session | -0.2 (0.86) | -0.2 (0.71) | -0.1 (0.83)
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.712, ANCOVA; GLM model with baseline as a covariate
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.607, ANCOVA; GLM model with baseline as a covariate

4. Secondary Outcome: Change in the Hypotension-induced Symptom Severity Score
Description: The hypotension-induced symptom severity score is the sum of a 6 question scale (each rated 0 [asymptomatic] to 4 [severe]). The questions look at cramps, dizziness, headache, nausea, itchiness, and restless legs syndrome experienced during dialysis.
  The outcome looks at the difference between the average baseline score (visits 2-7) and the average on-treatment scores (visits 14-19). The baseline value will be the arithmetic average of the values collected at each of the six baseline visits (visits 2-7). The on treatment value will be defined as the average of the values collected at each of the last six treatment visits (visits 14-19).
Time Frame: 6 weeks
Population: Patients must have completed visits in the visit 14-19 time frame.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 28 | 30 | 23
units on a scale | -0.9 (0.92) | -1.2 (1.32) | -1.2 (1.79)
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.4602, ANCOVA; GLM model with baseline as a covariate
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.940, ANCOVA; GLM model with baseline as a covariate

5. Secondary Outcome: Daily Symptoms Associated With Hemodialysis
Description: The Daily symptoms associated with hemodialysis score is the sum of an 8 question scale (each rated 0 [asymptomatic] to 4 [severe]). The questions look at fatigability, malaise/weakness, physical disturbance on standing, coldness of limbs, dizziness/lightheadedness, dizziness on standing, general bad feeling, and sleep disorders and asks how each of these items affected the patients daily activities on that day.
  The outcome looks at the difference between the average baseline score (visits 2-7) and the average on-treatment scores (visits 14-19). The baseline value will be the arithmetic average of the values collected at each of the six baseline visits (visits 2-7). The on treatment value will be defined as the average of the values collected at each of the last six treatment visits (visits 14-19).
Time Frame: 6 weeks
Population: Patients must have completed visits in the visit 14-19 timeframe. Three placebo patients and one droxidopa 600mg patient did not complete their Daily Symptoms Assessments during these visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 28 | 29 | 20
units on a scale | -0.13 (3.843) | -1.33 (3.724) | -1.34 (3.504)
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.376, ANCOVA; GLM model with baseline as a covariate
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.903, ANCOVA; GLM model with baseline as a covariate

6. Secondary Outcome: Change in the Multidimensional Fatigue Inventory (MFI-20)
Description: Fatigue will be measured by the general fatigue domain (items 1, 5, 12 and 16) of MFI-20 and will be summarized by treatment group and treatment period. The scores per item run from 1 to 5. A higher score indicates more fatigue. Therefore, the items indicative for fatigue need to be recoded (1=5, 2=4, 3=3, 4=2, 5=1). This concerns item: 5 and 16. A total score is calculated by summation of the scores of the individual items. Scores can range from the minimum of 4 to the maximum of 20.
  The value at baseline (visit 7) will be subtracted from the value on treatment (visit 19 or visit 13 if visit 19 is not available).
Time Frame: 6 weeks
Population: Patients must have completed at least visit 14. Three placebo patients did not complete their Multidimensional Fatigue Inventory during this visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 29 | 30 | 20
units on a scale | -0.1 (4.22) | -0.3 (2.93) | 0.6 (2.87)
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.319, ANCOVA; GLM model with baseline as a covariate
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.408, ANCOVA; GLM model with baseline as a covariate

7. Post Hoc Outcome: Systolic Blood Pressure Difference Between Pre-Hemodialysis and Nadir
Description: Change from baseline to end of study (HD visits 14-19) in systolic blood pressure difference between pre-hemodialysis and nadir.
Time Frame: 6 weeks
Population: Patients must have completed visits in the visit 14-19 timeframe. One droxidopa 400 mg patient did not have the required nadir blood pressure information for visits 14-19 and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 27 | 30 | 23
mmHg | -5.88 (13.638) | -3.33 (11.666) | 4.92 (18.180)
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA; GLM model with baseline as a covariate
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.030, ANCOVA; GLM model with baseline as a covariate

8. Other Pre Specified Outcome: Change in Systolic Blood Pressure From Pre-dialysis to Post-dialysis
Description: Change from baseline (visits 2-7) to end of study (HD visits 14-19) in the drop in systolic blood pressure from pre-hemodialysis to 5 minutes post-hemodialysis.
  The baseline value was the arithmetic average of the values collected at each of the six baseline visits (visits 2-7). The on treatment value was defined as the average of the values collected at each of the last six treatment visits (visits 14-19).
Time Frame: 6 weeks
Population: Patients must have completed visits in the visit 14-19 timeframe.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 28 | 30 | 23
mmHg | 3.41 (13.112) | 4.77 (11.556) | -4.39 (17.860)
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.025, ANCOVA; GLM model with baseline as a covariate
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.022, ANCOVA; GLM model with baseline as a covariate

9. Post Hoc Outcome: Number Patients With Hypotension Induced Early Termination of Dialysis Procedure
Time Frame: 6 weeks
Population: Patients had to have at least one post baseline visit (visit 8 and beyond).
Measure: Number; unit: participants
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Number analyzed (Participants) | 30 | 31 | 23
participants | 3 | 1 | 7
Statistical Analysis 1: Comparison: Droxidopa 400mg vs Placebo; Test type: Superiority or Other; p = 0.082, Fisher Exact
Statistical Analysis 2: Comparison: Droxidopa 600mg vs Placebo; Test type: Superiority or Other; p = 0.008, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Droxidopa 400mg | Droxidopa 600mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/30 | 5/31 | 6/23
Other Adverse Events (participants affected / at risk) | 20/30 | 18/31 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa 400mg (N=30) | Droxidopa 600mg (N=31) | Placebo (N=23)
Renal Transplane (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter Sepsis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Uremia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis Ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Indwelling Catheter Management (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Humerous Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Peripheral Artery Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa 400mg (N=30) | Droxidopa 600mg (N=31) | Placebo (N=23)
Procedural Nausea (Gastrointestinal disorders) | 5 (6) | 6 (9) | 3 (5)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2)
Asthenia (General disorders) | 4 (4) | 4 (4) | 2 (2)
Fatigue (General disorders) | 4 (4) | 6 (7) | 2 (2)
Feeling Abnormal (General disorders) | 4 (4) | 3 (3) | 2 (2)
Malaise (General disorders) | 4 (4) | 4 (4) | 1 (2)
Post Procedural Discomfort (General disorders) | 4 (4) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (3) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 (8) | 4 (6) | 2 (2)
Dizziness (Nervous system disorders) | 6 (7) | 3 (3) | 2 (3)
Dizziness Postural (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 5 (7) | 2 (2)
Poor Quality Sleep (Nervous system disorders) | 6 (7) | 4 (6) | 1 (1)
Restless Leg Syndrome (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days